CLINICAL TRIAL: NCT02468310
Title: Evaluating the Effects of Clinical Decision Making Support Systems on Maternal and Neonatal Mortality and Morbidity in Ghana: a Cluster Randomized Controlled Trial
Brief Title: Evaluating the Effects of SMS Text Messaging Support System Among Frontline Health Workers in Ghana
Acronym: Accelerate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannah Brown Amoakoh (Other)
Collaborators: Ghana Health Services (Other Government); University of Ghana (Other)
Responsible Party: Sponsor-Investigator, Hannah Brown Amoakoh, Clinical trials coordinator, Julius Global Health
Organization: Julius Global Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GHS-ERC: 10/09/14
Record Dates: First submitted 2015-06-07; First posted 2015-06-10 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Maternal Death; Neonatal Death; Postpartum Haemorrhage; Pre-eclampsia; Eclampsia; Pregnancy Induced Hypertension; Puerperal Sepsis; Asphyxia; Neonatal Sepsis; Neonatal Jaundice
Keywords: Maternal mortality; Neonatal mortality; Neonatal morbidity; Text messaging; Clinical decision making; Maternal Morbidity
MeSH Terms: conditions — Maternal Death; Perinatal Death; Postpartum Hemorrhage; Pre-Eclampsia; Eclampsia; Hypertension, Pregnancy-Induced; Puerperal Infection; Asphyxia; Neonatal Sepsis; Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention districts (Experimental): Access to protocols for management of obstetric and neonatal emergencies via text messaging on request in Intervention districts. Maternal and Neonatal emergency protocols
  Interventions: Other: Maternal and neonatal emergency protocols
- Control districts (No Intervention): No access to protocols for management of obstetric and neonatal emergencies via text messaging in control district

INTERVENTIONS:
Other: Maternal and neonatal emergency protocols — Protocols for management of Maternal and Neonatal emergencies based on the Safe Motherhood protocol adopted by the Ghana Health Service to improve maternal and neonatal health
  Other Names: Protocols for Maternal and Neonatal emergencies
  Arms: Intervention districts

SUMMARY:
Introduction Maternal and neonatal mortality continue to be to be prominent public health issues in sub Saharan Africa including Ghana, with slow progress made towards attainment of Millennium Development Goals (MDG) 4 & 5. Studies have identified poor quality of maternal and child healthcare as a major challenge to the prevention of neonatal and maternal deaths. Effective interventions are required to make significant inroads in these areas.

Objective To evaluate the effect of a SMS text messaging intervention to support clinical decision making by frontline health care professionals on neonatal and maternal mortality.

Methods We propose to conduct a randomized controlled trial in the Eastern region of Ghana, involving 8 intervention and 8 control districts. The intervention consists of text messaging of standard protocols for maternal and neonatal care to front line health care providers in the region. A total of 17,040 pregnant women who are receiving care (including antenatal, delivery and post-natal) at any of the hospitals in the selected districts in the region will be monitored through monthly aggregate data on outcome measures such as neonatal and maternal deaths from eclampsia, postpartum haemorrhage, puerperal sepsis, birth asphyxia, low birth weight and neonatal sepsis. Cord sepsis will also be included as neonatal sepsis for this study. Also, a quality of care assessment in four sampled districts to measure adherence to the safe motherhood protocol will be conducted. Stata software package.55 and MLwiN software version 2.2456 will be employed in data analysis. Descriptive analysis will be carried out to explore baseline characteristics of study groups while logistic regression will be applied to evaluate the effect of the intervention. A two-tailed statistical significant level of 0.05 will be used.

Expected outcome We hypothesize that the intervention will improve both maternal and neonatal service delivery and health outcomes in the intervention areas.

DETAILED DESCRIPTION:
Rationale of Study Based on the preponderance of evidence provided so far, Ghana is not on track for MDG 4 & 5.31 Despite increased antenatal care attendance in the health facilities,and the number of pregnancy delivered by skilled health care workers,neonatal and maternal mortality have not seen the needed decline.

Maternal deaths and neonatal deaths are caused by a complex interaction of economic, financial, social, cultural and clinical factors. Clinical factors are related to access to and quality of antenatal care, skilled attendance at delivery and emergency obstetric care. With over 90% of pregnant women receiving antenatal care from a health professional,it is believed that if adequate care is offered to these women, birth outcomes will be improved. Gaps identified in the quality of care given to pregnant women include poor quality of clinical decision guiding provider decisions on management choices.

Considering this we propose an evidence-based intervention facilitating easy access to maternal and neonatal guidelines for routine and emergency obstetric and antenatal/neonatal care for frontline providers, in public facilities. For the purpose of this intervention, we have chosen as a reference guideline the national Safe Motherhood protocol,an elaborate tool, that provides detailed state-of-the-art guidelines for maternal and newborn care, starting from prenatal care, through antenatal, delivery, postpartum, and newborn care. We chose text messaging based on the Unstructured Supplementary Service Data (USSD) system as a low-cost, easily-accessible and instant way of requesting needed information in standard and emergency situations by the health care provider to enhance clinical decision making.

Objectives Primary objective

* To assess the quantitative effect of USSD-based text messaging of standard protocols for maternal and neonatal care on the incidence of neonatal mortality Secondary objectives
* To assess the quantitative effect of USSD-based text messaging of standard protocols for maternal and neonatal care on the incidence of maternal mortality
* To assess the quantitative effect of USSD-based text messaging of standard protocols for maternal and neonatal care on the incidence of neonatal morbidity
* To assess the quantitative effect of USSD-based text messaging of standard protocols for maternal and neonatal care on the incidence of maternal morbidity
* To assess adherence of health care providers to clinical guidelines for maternal antenatal care

Study design A cluster randomized controlled trial49 design will be used to examine the effect of CDMSS in the form of USSD-based text messaging of standard protocols for the management of maternal and neonatal care to providers, on neonatal and maternal mortality in the Eastern region, Ghana. This research is planned to commence in January 2015 and end in June 2016. Each of the districts in the region will be the cluster unit of randomization. This design was adopted in order to avoid contamination both at the patient and health professional levels, which may occur as a result of social interaction.

After randomization, a baseline study will be conducted in the districts and facilities to collect data on district and facility characteristics, while baseline measures of the chosen outcomes will be obtained from the District Health Information Management System - 2 (DHIMS - 2) which has been shown to provide accurate estimates of neonatal health indicators.50 This will take place from November to December 2014. The baseline study will be followed by the intervention study that will run for a period of 18 months. During this period monthly monitoring, including data collection of the outcome measures will be carried out by the study team. In addition, a quality of care study, done by assessment of provider adherence to the guidelines sent through the SMS text messaging will be conducted in 2 selected districts each from the intervention and control districts, through a record review of a random sample of clients seen during the period. The process of implementation of the intervention will be documented. At the end of the intervention period, a post intervention evaluation will be carried out at the district and facility level.

ELIGIBILITY:
Inclusion Criteria:

* District location in the Eastern region of Ghana.
* The districts should have an expected deliveries of ≥ 1,100 / year
* The District Health Management Team and the District Hospital Management Team must agree to participate in the study.

Exclusion Criteria:

* District location outside the Eastern region.
* The districts expected deliveries of <1,100 / year
* The District Health Management Team and the District Hospital Management Team disagreeing to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65831 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-04-09 (Actual)

PRIMARY OUTCOMES:
Number of neonatal deaths | 18 months
  Total number of neonatal deaths among total number of deliveries over an 18 month period

SECONDARY OUTCOMES:
Number of maternal deaths | 18 months
  Total number of maternal deaths among total antenatal attendants over an 18 month period
Number of cases of eclampsia | 18 months
  Total number of cases of eclampsia among total antenatal attendants over an 18 month period
Number of cases of postpartum haemorrhage | 18 months
  Total number of cases of postpartum haemorrhage among total antenatal attendants over an 18 month period
Number of cases of prolonged labour | 18 months
  Total number of cases of prolonged labour among total antenatal attendants over an 18 month period
Number of cases of puerperal sepsis | 18 months
  Total number of cases of puerperal sepsis among total antenatal attendants over an 18 month period
Number of cases of birth asphyxia among deliveries | 18 months
  Total number of cases of birth asphyxia among total deliveries over an 18 month period
Number of cases of low birth weight deliveries | 18 months
  Total number of cases of low birth deliveries among total deliveries over an 18 month period
Number of cases of cord sepsis | 18 months
  Total number of cases of cord sepsis among total deliveries over an 18 month period

OTHER OUTCOMES:
Percentage of cases of pre-eclampsia/Pregnancy induced hypertension appropriately managed | 18 months
  This will measure the percentage of cases of pre-eclampsia/pregnancy induced hypertension managed according to the Safe Motherhood Protocol
Percentage of cases of birth asphyxia appropriately managed | 18 months
  This will measure the percentage of cases of birth asphyxia managed according to the Safe Motherhood Protocol

CONTACTS AND LOCATIONS:
Overall Officials: Irene Agyepong, MD DRPH PhD, Principal Investigator — Julius Center University of Utrecht
Locations (1):
- Eastern Region Health directorate, Koforidua, Ghana

IPD SHARING:
Plan to Share IPD: Undecided
Permission needs to be sought from Ghanaian health authorities first.

REFERENCES:
- [Derived] Amoakoh HB, Klipstein-Grobusch K, Agyepong IA, Zuithoff NPA, Amoakoh-Coleman M, Kayode GA, Sarpong C, Reitsma JB, Grobbee DE, Ansah EK. The effect of an mHealth clinical decision-making support system on neonatal mortality in a low resource setting: A cluster-randomized controlled trial. EClinicalMedicine. 2019 Jul 4;12:31-42. doi: 10.1016/j.eclinm.2019.05.010. eCollection 2019 Jul. PMID 31388661
- [Derived] Amoakoh HB, Klipstein-Grobusch K, Amoakoh-Coleman M, Agyepong IA, Kayode GA, Sarpong C, Grobbee DE, Ansah EK. The effect of a clinical decision-making mHealth support system on maternal and neonatal mortality and morbidity in Ghana: study protocol for a cluster randomized controlled trial. Trials. 2017 Apr 4;18(1):157. doi: 10.1186/s13063-017-1897-4. PMID 28372580